CLINICAL TRIAL: NCT02990455
Title: Reduced Nicotine Cigarettes in Smokers With and Without Alcohol Use Disorder
Acronym: RedNic
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Battelle Memorial Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: BMI-202181
Record Dates: First submitted 2016-12-07; First posted 2016-12-13 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Alcohol Drinking; Cigarette Smoking Toxicity
Keywords: alcohol; drinking; smoking; cigarette; nicotine
MeSH Terms: conditions — Alcohol Drinking; Smoking

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduced Nicotine Cigarette - Moderate (Experimental): Nicotine Research Cigarette Drug Supply Program Category Codes NRC600 and NRC601 (menthol); each cigarette contains 0.8mg nicotine; participants will be instructed to smoke these cigarettes according to their usual smoking patterns
  Interventions: Drug: Reduced nicotine cigarettes
- Reduced Nicotine Cigarette - Low (Experimental): Nicotine Research Cigarette Drug Supply Program Category Codes NRC102 and NRC103 (menthol); each cigarette contains 0.03mg nicotine; participants will be instructed to smoke these cigarettes according to their usual smoking patterns
  Interventions: Drug: Reduced nicotine cigarettes

INTERVENTIONS:
Drug: Reduced nicotine cigarettes — Participants will be assigned to undergo two experimental conditions (i.e., exclusive smoking of RNC Low or Moderate in their home environment for 7 days) in a double-blind, randomized, crossover design. The two experimental conditions will be separated by a 7-day period of return to smoking of participants' own brand of cigarette.
  Other Names: Nicotine research cigarettes

SUMMARY:
The proposed research will investigate whether smokers with vs. without current at-risk alcohol drinking (ARD) respond to reduced nicotine cigarettes by increasing their alcohol consumption or smoke exposure, thereby diminishing the hypothesized public health benefit of these new products.

DETAILED DESCRIPTION:
The current proposal examines response to two RNCs, one with low nicotine content (RNC Low; 0.03mg) and one with moderate nicotine content (RNC Moderate; 0.8mg) in daily smokers with and without ARD. Participants (N = 70) will attend a total of five visits to the laboratory. The first visit will be to classify participants as either ARD (n = 35) or Non ARD (n = 35) and gather baseline data. Participants will be assigned to undergo two experimental conditions (i.e., exclusive smoking of RNC Low or Moderate in their home environment for 7 days) in a double-blind, randomized, crossover design. The two experimental conditions will be separated by a 7-day period of return to smoking of participants' own brand of cigarette. On the first and last day of each of the two experimental conditions, participants will smoke the assigned RNC in the laboratory, and data on toxicant exposure (i.e., boost in exhaled carbon monoxide and plasma nicotine and cotinine; solanesol from smoked cigarette butts), subjective acceptability (i.e., subjective response; risk perceptions; relative reinforcing efficacy); and smoking compensation (i.e., smoking topography measures) related to the smoked RNC will be collected. During each 7-day period of exposure to the RNCs, participants will provide daily data on alcohol and nicotine use, nicotine withdrawal, smoking urge, and alcohol urge via telephone-based Interactive Voice Response technology. The strength of our study design is that we can evaluate both between-group (i.e., ARD vs. Non ARD) and within-person (i.e., RNC Low vs. Moderate) differences in response to RNCs and, furthermore, can examine whether increased nicotine withdrawal, smoking urge, and alcohol urge mediate the relation between decreased nicotine exposure and alcohol consumption. Results from this study will show what mechanisms underlying drinking and smoking may need to be addressed in future integrated interventions for both problems and will immediately inform the practical implementation of market-wide reductions in cigarette nicotine content among smokers with ARD.

ELIGIBILITY:
Inclusion Criteria:

* Ages 21-65;
* Smokes ≥ 10 cigarettes/day for ≥ 2 years;
* Has no immediate plans to quit drinking or smoking; and
* Sufficient understanding of informed consent form and study procedures.

Exclusion Criteria:

* Has or is at-risk of serious alcohol-related consequences, defined as any of the following:

  1. Meets DSM-5 criteria for current alcohol use disorder with the presence of 6 or more symptoms (i.e., current severity of severe)
  2. Has a Clinical Institute Withdrawal Assessment scale score of ≥8,
  3. Self-report of history of seizures, delirium, or hallucinations during alcohol withdrawal;
  4. Self-report of drinking to avoid withdrawal symptoms, or
  5. Self-report of a history of alcohol withdrawal treatment.
* Women if pregnant, lactating, or not using a reliable form of birth control;
* Has current serious psychiatric disorder;
* Has DSM-5 current severe substance use disorder, other than nicotine;
* Has current use of smokeless tobacco, pipes, cigars, e-cigarettes, or nicotine replacement products;
* Displays clinically evident intoxication on any study visit, confirmed by breathalyzer test (breath alcohol level (BAL)>0.02 mg%);
* Has difficulties with blood draws or poor venous access; or
* Has significant smoking-related disease (by history).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-04-21 (Actual)

PRIMARY OUTCOMES:
Alcohol drinks per day | 7 days

SECONDARY OUTCOMES:
Toxicant exposure | 7 days
  (1) boost in (a) exhaled carbon monoxide, (b) plasma nicotine, and (c) plasma cotinine, and (2) solanesol after laboratory smoking
Subjective acceptability | 7 days
  subjective response
Smoking compensation | 7 days
  number of cigarettes per day during each 7-day period

CONTACTS AND LOCATIONS:
Locations (1):
- Battelle Memorial Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No